CLINICAL TRIAL: NCT05552300
Title: Effectiveness and Safety of Superselective Adrenal Arterial Embolization (SAAE) for Resistant Hypertension: A Randomized, Parallel, Controlled Clinical Trial
Brief Title: Superselective Adrenal Arterial Embolization for Resistant Hypertension
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: First Affiliated Hospital of Chengdu Medical College (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SAAE-RHT
Record Dates: First submitted 2022-09-11; First posted 2022-09-23 (Actual); Last update posted 2022-09-23 (Actual); Status verified 2022-09

CONDITIONS: Resistant Hypertension

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Superselective adrenal arterial embolization (Experimental): Selectively injects ethanol into adrenal artery to ablate part of the adrenal gland
  Interventions:
  Procedure: superselective adrenal arterial embolization Drug: traditional triple antihypertensive treatment
  Interventions: Procedure: SAAE; Drug: traditional triple antihypertensive treatment
- Traditional triple antihypertensive treatment (Active Comparator): No intervention, but treated with traditional triple antihypertensive treatment
  Interventions: Drug: traditional triple antihypertensive treatment

INTERVENTIONS:
Procedure: SAAE — SAAE is a catheter-based percutaneous transluminal procedure which selectively injects ethanol into adrenal artery to ablate part of the adrenal gland for suppression of excessive aldosterone and catecholamines
  Arms: Superselective adrenal arterial embolization
Drug: traditional triple antihypertensive treatment — irbesartanhydrochlorothiazide 162.5 mg/d, amlodipine 5 mg/d

SUMMARY:
Resistant hypertension (RH) is usually defined as blood pressure (BP) that remains above guideline-specified targets despite the use of three or more antihypertensive agents at optimal or maximally tolerated doses, with one of those agents preferably being a diuretic. It is not uncommon, being identified in 10 to 30% of hypertensive patients and it is known to be a risk factor for cardiovascular (CV) events, including stroke, myocardial infarction (MI), heart failure (HF), and CV mortality, as well as adverse renal events,including chronic kidney disease (CKD) and end-stage kidney disease (ESKD). The activation of the renin-angiotensin-aldosterone system (RAAS) and sympatho-adrenomedullary system can play a pathogenic role in triggering and sustaining RH. SAAE is a catheter-based percutaneous transluminal procedure which selectively injects ethanol into adrenal artery to ablate part of the adrenal gland for suppression of excessive aldosterone and catecholamines. Therefore, SAAE is a minimally invasive procedure that might be used as an alternative strategy to antihypertensive drugs or reduce the intensity of antihypertensive drugs.

DETAILED DESCRIPTION:
Not Provided

ELIGIBILITY:
Inclusion Criteria:

* Male or female, aged between 18-65 years old.
* Patients with resist hypertension (office systolic blood pressure ≥140 mmHg, and/or office diastolic blood pressure ≥90 mmHg, and/or 24-h average systolic blood pressure ≥130 mmHg) with rational lifestyle change and triple antihypertensive drugs (irbesartanhydrochlorothiazide 162.5 mg/d, amlodipine 5 mg/d) for at least 4 weeks.
* Informed consent signed and agreed to participate in this trial.

Exclusion Criteria:

* Secondary hypertension
* Adrenergic insufficiency.
* adrenocortical insufficiency
* Renal failure eGFR<60 mL/min/1.73 m2
* Heart failure with NYHA grade Ⅱ-Ⅳ grade or unstable angina, severe cardiovascular and cerebrovascular stenosis, myocardial infarction, intracranial aneurysm, stroke and other acute cardiovascular events.
* Acute infections, tumors and severe arrhythmias, psychiatric disorders, drugs or alcohol addicts.
* Liver dysfunction or the following history of liver disease: AST or ALT 3 times higher than the upper limit, liver cirrhosis, history of hepatic encephalopathy, esophageal variceal history or portal shunt history.
* Fertile woman without contraceptives.
* Coagulation dysfunction.
* Pregnant women or lactating women.
* Participated in other clinical trials or admitted with other research drugs within 3 months prior to the trial.
* Any surgical or medical condition which can significantly alter the absorption, distribution, metabolism, or excretion of any study drug.
* Allergy or any contraindications for the study drugs, contrast agents and alcohol.
* History of depression, schizophrenia or vascular dementia.
* Refused to sign informed consent

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 144 (Estimated)
Dates: Start 2022-10-01 (Estimated); Primary Completion 2024-10-01 (Estimated); Study Completion 2025-03-31 (Estimated)

PRIMARY OUTCOMES:
Change of 24-h average systolic blood pressure | 6-month
  Difference in the change of 24-h average systolic blood pressure between the intervention and control group

SECONDARY OUTCOMES:
Change of 24-h average diastolic blood pressure, daytime mean systolic blood pressure, daytime mean diastolic blood pressure, and nighttime average systolic and diastolic blood pressure | 6-month
  Difference in the change of 24-h average diastolic blood pressure, daytime mean systolic blood pressure, daytime mean diastolic blood pressure, and nighttime average systolic and diastolic blood pressure between the intervention and control group
Change of the number of antihypertensive medications | 6-month
  Difference in the change of the number of antihypertensive medications between the intervention and control group
Change of home systolic and diastolic pressure | 6-month
  Difference in the change of home systolic and diastolic pressure between the intervention and control group
Change of office systolic and diastolic pressure | 6-month
  Difference in the change of office systolic and diastolic pressure between the intervention and control group
Change of blood electrolytes (K+, Na +) | 6-month
  Difference in the change of blood electrolytes (K+, Na + in mmol/L) between the intervention and control group
Change of plasma aldosterone | 6-month
  Difference in the change of plasma aldosterone (pg/mL) between the intervention and control group
Change of plasma cortisol | 6-month
  Difference in the change of plasma cortisol (nmol/L) between the intervention and control group
Change of plasma renin measured | 6-month
  Difference in the change of plasma renin (pg/ml) between the intervention and control group
Change of liver enzymes | 6-month
  Difference in the change of liver enzymes (ALT, AST in IU/L) between the intervention and control group
Change of kidney function | 6-month
  Difference in the change of serum creatinine in umol/L between the intervention and control group
Change of fasting blood glucose | 6-month
  Difference in the change of fasting blood glucose in mmol/L between the intervention and control group
Change of lipids profiles | 6-month
  Difference in the change of lipids profiles (TC, HDL-C, LDL-C, TG) in mmol/L between the intervention and control group
Change of 24-h urine microalbumin | 6-month
  Difference in the change of 24-h urine microalbumin (mg/L) between the intervention and control group
Change of 24-h 24-h urine creatinine | 6-month
  Difference in the change of 24-h urine creatinine (umol/L) between the intervention and control group
Change of echocardiography parameters (LVEF) | 6-month
  Difference in the change of cardiac parameters assessed by echocardiography LVEF (%) between the intervention and control group
Change of echocardiography parameters (IVSd、IVSs、LVPWd, LVPWs, LVEDD) | 6-month
  Difference in the change of echocardiography parameters (IVSd、IVSs、LVPWd, LVPWs, LVEDD, in millimetre[mm]) between the intervention and control group
Change of carotid intima-media thickness | 6-month
  Difference in the change of carotid intima-media thickness(CIMT) assessed by carotid ultrasound between the intervention and control group

CONTACTS AND LOCATIONS:
Overall Officials: Peijian Wang, Study Chair — Clinical Medical College and The First Affiliated Hospital of Chengdu Medical College

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Bourque G, Hiremath S. Rethinking Resistant Hypertension. J Clin Med. 2022 Mar 7;11(5):1455. doi: 10.3390/jcm11051455. PMID 35268545
- [Result] Dong H, Zou Y, He J, Deng Y, Chen Y, Song L, Xu B, Gao R, Jiang X. Superselective adrenal arterial embolization for idiopathic hyperaldosteronism: 12-month results from a proof-of-principle trial. Catheter Cardiovasc Interv. 2021 May 1;97 Suppl 2:976-981. doi: 10.1002/ccd.29554. Epub 2021 Feb 19. PMID 33605538
- [Result] Giurazza F, Corvino F, Silvestre M, Cangiano G, Cavaglia E, Amodio F, De Magistris G, Frauenfelder G, Niola R. Adrenal glands hemorrhages: embolization in acute setting. Gland Surg. 2019 Apr;8(2):115-122. doi: 10.21037/gs.2018.10.06. PMID 31183321
- [Result] Zhou Q, Liu X, Zhang H, Zhao Z, Li Q, He H, Zhu Z, Yan Z. Adrenal Artery Ablation for the Treatment of Hypercortisolism Based on Adrenal Venous Sampling: A Potential Therapeutic Strategy. Diabetes Metab Syndr Obes. 2020 Oct 6;13:3519-3525. doi: 10.2147/DMSO.S262092. eCollection 2020. PMID 33116703
- [Result] Zhao Z, Liu X, Zhang H, Li Q, He H, Yan Z, Sun F, Li Y, Zhou X, Bu X, Wu H, Shen R, Zheng H, Yang G, Zhu Z; Chongqing Endocrine Hypertension Collaborative Team. Catheter-Based Adrenal Ablation Remits Primary Aldosteronism: A Randomized Medication-Controlled Trial. Circulation. 2021 Aug 17;144(7):580-582. doi: 10.1161/CIRCULATIONAHA.121.054318. Epub 2021 Aug 16. No abstract available. PMID 34398686